CLINICAL TRIAL: NCT05109780
Title: Feasibility of "EmoGuía" to Guide and Personalize Psychological Treatments
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitat Jaume I (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: EMIUJI
Record Dates: First submitted 2021-09-27; First posted 2021-11-05 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-02

CONDITIONS: Emotional Disorder
Keywords: My EMI, Emotional Wellbeing; Transdiagnostic approach; Emotional Disorder; Unified Protocol

STUDY DESIGN:
Intervention Model Description: One condition
Masking Description: Patients will be informed of the condition they have been assigned to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- App + Unified Protocol Arm (Experimental): Participants at this condition will be daily monitored by the app (My Emi, Emotional Well-being) while they are administered a self-applied online transdiagnostic intervention for their emotional disorders. Alarms will be generated in the face of certain pre-set undesired events.
  Therapists will receive pre-set clinical alarms in real time in the presence of relevant clinical events previously determined by the clinical staff (e.g., clinical worsening or no improvement of functionality, mood or psychological mechanisms worked in therapy). This information will be used to make clinical decisions in a short period of time (e.g., call the patient, or send additional therapeutic material by mail or through the app (momentary ecological intervention), or for its implementation during the course of psychological therapy in order to make the therapy more efficient, safe, personalized and adapted to the needs of the patient.
  Interventions: Device: My EMI, Emotional Well-being + self-applied online transdiagnostic treatment

INTERVENTIONS:
Device: My EMI, Emotional Well-being + self-applied online transdiagnostic treatment — The intervention will consist in a self-applied online transdiagnostic intervention for emotional problems together with an app-based EMI. In terms of monitoring, the My EMI, Emotional Well-being is a mobile app whose contents have been adapted to conduct ecological momentary assessments in different health conditions. The app assesses important psychological variables, namely anxiety, depressive symptoms,etc. Participants respond daily to the questions in the app. In terms of the online self-applied intervention, the Unified Protocol is a transdiagnostic extension of CBT which works on regulate emotions in a more adaptive way through 5 core treatment modules: present-focused emotional awareness, cognitive flexibility, identification and prevention of emotional avoidance patterns, increasing awareness and tolerance to emotion-elicited physical sensations, and graded (interoceptive and situational) exposure procedures.
  Other Names: My EMI, Emotional Well-being

SUMMARY:
The present project aims at testing the feasibility of an app-based system called "EmoGuía" for routine outcome monitoring of adult patients with emotional disorders while they are administered a self-applied online transdiagnostic psychological intervention.

DETAILED DESCRIPTION:
Anxiety and depressive disorders, commonly known as emotional disorders (EDs), are the most frequent mental health problems why patients seek for medical care globally. According to recent epidemiologic studies, lifetime prevalence rates reveal that anxiety and depression disorders affect approximately an estimated 31.9% and 33.7% of people worldwide, respectively. In Spain, a nationwide study showed a prevalence of anxiety and depression disorders of 5.2% and 4.1%, approximately. Consequently, EDs lead to considerable direct and indirect economic losses for countries, as well as a great negative impact on the quality of life and overall functioning of individuals. Adding up to the previous, the current covid-19 pandemic not only has boosted the incidence of mental disorders in healthy people, but also has exacerbated emotional problems in vulnerable populations.

Encouragingly, the effectiveness of psychotherapy for the treatment of EDs, especially cognitive behavioural therapy (CBT), has been supported by a vast amount of scientific evidence. In particular, Internet-delivered CBT (iCBT), where patients sign in to a safe website to access online psychotherapeutic materials within several modules, has emerged in recent years as an effective alternative to face-to-face psychotherapy in an attempt to reduce costs, save therapists' and clients' time, bring psychological treatments closer to the population, and disseminate interventions easily. The growth of digital care has become even more obvious during the covid-19 pandemic and the associated quarantine, where great efforts have been made to adapt evidence-based treatments to a new digital format. Therefore, the current situation has become an opportunity to develop and implement promising digital interventions, which are now more sensible than ever.

To make evidence-based treatments even more accessible, extensions and innovations of CBT have been developed in recent years. The latest research supports a transdiagnostic perspective for the treatment of EDs, where cognitive-behavioural techniques are included to target different EDs altogether. Indeed, the transdiagnostic approach appears to be an effective alternative to single disorder interventions in order to address the high comorbidity rates between anxiety and depressive disorders, as well as the shared mechanisms and the overlapping symptomatology across different disorders which play an essential role in the onset and maintenance of them. In particular, the Unified Protocol (UP), a transdiagnostic extension of CBT which works on regulate emotions in a more adaptive way through different core treatment modules, has been developed for the treatment of EDs. Specifically, the UP shows promising effects not only when delivered onsite, but also online, which makes it an excellent psychological approach to reach a large number of individuals with a single treatment protocol.

In this line, some interesting proposals emphasize the need for a paradigm shift from randomized controlled trials that work on average towards personalized treatments that allow to focus more on the individual (to avoid what group average can mask). In particular, measurement-based care, which consists of routine patient monitoring, periodic feedback to the therapist (or both therapist and patient), and adaptation of the intervention according to such feedback appears to be a feasible option in order to adapt treatments to patients' needs. Fortunately, with the rapid growth of new technologies in our society such as mobile applications (apps), measurement-based care can be implemented more effectively as the apps can be used as support tools for the assessment of several psychological outcome variables. This procedure is commonly known as Ecological Momentary Assessment (EMA) and can help overcome some of the obstacles that traditional, retrospective face-to-face assessments hold. EMA has the potential to assess patients repeatedly and frequently over time, allows to observe fluctuations in patient outcomes, and early interventions can be administered in response to pre-set clinical alarms.

To our knowledge, studies that use technology to improve the management of emotional problems have generally opted for using apps that report on the evolution of treatment to obtain more reliable measures of the evolution of patients or, more frequently, have used different technologies such as web pages or apps to facilitate self-applied treatments based on pre-established modules. The present study goes one step further and explores not only the usefulness of the EMA by means of an app for the improvement of the assessment process of patients with emotional problems/EDs, but also the feasibility of using it to make adjustments in real time or very short-term (e.g., in weekly visits) during the psychotherapeutic process, resembling an ecological momentary intervention (EMI). Several studies have supported the use of EMA to deliver the most personalized feedback or psychological support in real life for a given patient in order to enhance psychotherapy effectiveness and facilitate tailored treatments.

Objectives The current study aims to explore the feasibility of an app-based system called "EmoGuía" a recently developed app that will provide personalized measurement-based care (MBC) based on EMIs according to the patients' daily evolution observed with daily evolution/assessment observed in the app (Castilla et al., 2022a). The EMI app will complement a self-applied online transdiagnostic treatment for people with EDs, which has shown to be effective in past research (Díaz-García et al., 2021).

The objectives of this feasibility study are: (1) to test whether the EMI app is appraised as simple to use, useful and acceptable by both patients and psychologists (app usability, satisfaction, and acceptability) and, (2) to test the number of completed assessments and transdiagnostic modules from those suggested (adherence to the app and treatment compliance). As a secondary goal, we will investigate the potential effectiveness of the EMI app by exploring whether changes in outcome variables and mechanisms of change (anxiety, depression, and emotion regulation) occur after the app use at an individual level.

We anticipate that the implementation of the app "EmoGuía" will be feasible in terms of usability, satisfaction, acceptability, compliance, retention rates, and adherence. Thus, we expect that patients and psychologists will perceive the app to be useful, will experience low burden associated with its use, and will be satisfied with the procedure. We also expect to improve the mood status and emotion regulation outcomes in a large number of participants.

The design of a future clinical trial will be optimized with the aforementioned objectives. The current article describes the study protocol of this trial.

ELIGIBILITY:
Inclusion Criteria:

1. age ≥18 years
2. showing problematic levels (one standard deviation above or below the mean) in at least one of the 9 transdiagnostic dimensions of the Multidimensional Emotional Disorders Inventory (MEDI; Osma et al., 2021; Rosellini & Brown, 2019) or having moderate-to-severe anxiety (scores ≥8) or depressive symptoms (scores ≥5), as reported in the Overall Anxiety Severity and Impairment Scale (OASIS) and the Overall Depression Severity and Impairment Scale (ODSIS) (Mira et al., 2019)
3. having the ability to read and understand Spanish
4. having a computer and a mobile phone Internet access
5. signing the online informed consent.

Exclusion criteria:

1. age <18
2. severe mental health problems
3. high suicide risk
4. receiving psychological treatment for the same ED emotional problem targeted by our study at the same time the current study is being conducted
5. <8 in OASIS and <5 in ODSIS, or non-problematic scores in the MEDI
6. have changes and/or increases in pharmacological treatment during the study (stable medication will be accepted).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2024-03-01 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
App' usability and acceptability | It will be assessed at the end of the study, after 18 weeks
  My EMI, Emotional Well-being will be assessed by the System Usability Scale in order to evaluate the perception that this tool is simple to use and useful. It is composed by 10 items which are responded according to a 5-point Likert scale (1 = "completely disagree" to 5 ="completely agree").
Adherence to the app and treatment | One time once the study finishes, after 18 weeks
  Participants' adherence to the app (response rate) will be calculated by dividing the number of the completed assessments in the app by the number of planned evaluations (percentage of daily assessments completed from the assessments prompted). Additional data will be passively collected from the online treatment platform and the app. From the online treatment, the number of modules completed and the number of tasks completed in the online intervention will be collected.
App satisfaction | One time once the study finishes, after 18 weeks
  Satisfaction with the app and perceived burden will be evaluated using questions developed by our team and used in previous works using technology (Suso-Ribera, Castilla, Zaragozá, Ribera-Canudas, Botella, & García-Palacios, 2018). Example items will be "To what extent are you satisfied with the app?" and "To what extent would you recommend the app?".
Feasibility of the support call and videoconference | One time once the study finishes, after 18 weeks
  We will also record the number of support calls and videoconferences made as a function of the alarms received, the response rate by patients to this supportive care, and their duration.

SECONDARY OUTCOMES:
Overall Anxiety Severity and Impairment Scale | At the beginning of the study, at the end of the study (18 weeks after using the app) and 3 month follow-up
  It consists of 5 questions that measure the severity and interference of anxiety during the previous week (Osma et al., 2019). The total scale score ranges from 0 to 20. Items are rated on a 5-point Likert scale ranging from 0 to 4. The Spanish validation has shown excellent internal consistency estimates (Cronbach's alpha was 0.87) in patients with EDs (Osma et al., 2019).
Overall Depression Severity and Impairment Scale | At the beginning, at the end of the study (18 weeks after using the app) and 3 month follow-up
  It consists of 5 questions that measure the severity and interference of depression during the previous week (Osma et al., 2019). Again, the total scale score ranges from 0 to 20. Items are rated on a 5-point Likert scale ranging from 0 to 4. The Spanish validation has shown excellent internal consistency estimates (Cronbach's alpha was 0.94) in patients with EDs (Osma et al., 2019).
Multidimensional Emotional Disorders Inventory | At the beginning, at the end of the study (18 weeks after using the app) and 3 month follow-up
  The MEDI has 49 questions grouped in 9 dimensions (Osma et al., 2021). The Spanish validation of the MEDI has shown excellent reliability indices as estimated with the internal consistency of the nine factors (Cronbach's alphas between 0.74 and 92) (Osma et al., 2021).
EMAs | Daily monitoring (10 days before the intervention begins and during treatment)
  Outcome variables (anxiety, depression, anger, happiness, activity level) and mechanisms of change (understanding role of emotions, mindfulness, cognitive flexibility, Emotional avoidance, Tolerance to unpleasant physical sensations, and Behaviours not guided by emotion)

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Gual- Montolio, Study Chair — Universitat Jaume I; Juana Maria Bretón-López, Study Chair — Universitat Jaume I

IPD SHARING:
Plan to Share IPD: No
Individual Participant Data (IPD) will not be shared with other researchers.

REFERENCES:
- [Background] Suso-Ribera C, Castilla D, Zaragoza I, Ribera-Canudas MV, Botella C, Garcia-Palacios A. Validity, Reliability, Feasibility, and Usefulness of Pain Monitor: A Multidimensional Smartphone App for Daily Monitoring of Adults With Heterogenous Chronic Pain. Clin J Pain. 2018 Oct;34(10):900-908. doi: 10.1097/AJP.0000000000000618. PMID 29659375
- [Background] Barlow DH, Farchione TJ, Fairholme CP, Ellard KK, Boisseau CL, Allen LB, Ehrenreich-May J. Protocolo unificado para el tratamiento transdiagnóstico de los trastornos emocionales: Manual del terapeuta y manual del paciente. [The unified protocol for transdiagnostic treatment of emotional disorders: Client workbook and Therapist guide]. Madrid: Alianza Editorial; 2015.
- [Background] Osma J, Castellano C, Crespo E, García-PalaciosA. The Unified Protocol for Transdiagnostic Treatment of Emotional Disorders in format group in a Spanish public mental health setting. PsicologíaConductual. 2015; 23 (3): 447-466.
- [Background] Gual-Montolio P, Martinez-Borba V, Breton-Lopez JM, Osma J, Suso-Ribera C. How Are Information and Communication Technologies Supporting Routine Outcome Monitoring and Measurement-Based Care in Psychotherapy? A Systematic Review. Int J Environ Res Public Health. 2020 May 2;17(9):3170. doi: 10.3390/ijerph17093170. PMID 32370140
- [Background] Colombo D, Fernandez-Alvarez J, Suso-Ribera C, Cipresso P, Valev H, Leufkens T, Sas C, Garcia-Palacios A, Riva G, Botella C. The need for change: Understanding emotion regulation antecedents and consequences using ecological momentary assessment. Emotion. 2020 Feb;20(1):30-36. doi: 10.1037/emo0000671. PMID 31961174
- [Derived] Gual-Montolio P, Suso-Ribera C, Garcia-Palacios A, Castilla D, Zaragoza I, Breton-Lopez J. Enhancing Internet-based psychotherapy for adults with emotional disorders using ecological momentary assessments and interventions: Study protocol of a feasibility trial with "My EMI, Emotional Well-being" app. Internet Interv. 2023 Jan 5;31:100601. doi: 10.1016/j.invent.2023.100601. eCollection 2023 Mar. PMID 36686334